CLINICAL TRIAL: NCT06198257
Title: Comparative Effects of Spider Cage Therapy and Modified Suit Therapy on Trunk Stability and Pelvic Control in Children With Cerebral Palsy
Brief Title: Comparative Effects of Spider Cage Therapy and Modified Suit Therapy in CP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/RCR&AHS/23/0764
Record Dates: First submitted 2023-12-26; First posted 2024-01-10 (Actual); Last update posted 2024-06-13 (Actual); Status verified 2024-06

CONDITIONS: Cerebral Palsy
Keywords: CP; Pelvic control; Spider cage therapy; modified Thera suits
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Intervention Model Description: It will be Randomized Controlled trial in which non probability convenience sampling technique will be used. Two groups of 8 to 12 age will be formed in which participants will be randomly divided by lottery method. Group A will be given modified Thera suits and the other group B will receive spider cage therapy on trunk stability and pelvic control.
Who Masked: Participant
Masking Description: Participants will get seperate treatment protocols and possible efforts will be put to mask the both groups about their treatment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- group A (Active Comparator): Spider cage therapy along with strengthening exercises
  Interventions: Device: spider cage
- group B (Active Comparator): Modified suits therapy along with strengthening exercise
  Interventions: Device: modified suits therapy

INTERVENTIONS:
Device: spider cage — 5 days a week for an hour/daily with conventional exercises. Assisted sit to stand (10 to 15---15 to 20) Assisted weight shift (10 to 15---15 to 20) Assisted trunk rotation (10 to 15---15 to 20) Hip Abd / Add. exercises (10 to 15---15 to 20) Bridge exercises (10 to 15---15 to 20)
  Arms: group A
Device: modified suits therapy — 5 days a week for an hour/daily with conventional exercises. Assisted sit to stand (10 to 15---15 to 20) Assisted weight shift (10 to 15---15 to 20) Assisted trunk rotation (10 to 15---15 to 20) Hip Abd / Add. exercises (10 to 15---15 to 20) Bridge exercises (10 to 15---15 to 20)
  Arms: group B

SUMMARY:
Spider Cage is a part of universal exercise unit. It is a suspension system, which works with use of belts, elastic cords and Thera suits (Thera suits especially for cerebral palsy). Cords are dynamic and provides an appropriate amount of support with the help of which patient can perform movement independently. Cerebral Palsy (CP) is a condition where non progressive disorders of posture caused by abnormal development of, or damage to, motor control centers of brain resulting in abnormal movements.

DETAILED DESCRIPTION:
It will be Randomized Controlled trial in which non probability convenience sampling technique will be used. Two groups of 8 to 12 age will be formed in which participants will be randomly divided by lottery method. Group A will be given modified Thera suits and the other group B will receive spider cage therapy on trunk stability and pelvic control. Improvement will be identified by Trunk Control Measurement Scale (TCMS), Trunk impairment scale (TIS) and Gross motor function classification system. (GMFCS) level I-II. The result after statistical analysis will show that which treatment will be more effective. Results will be analyzed on SPSS 29. Data analyzed by repeated measures ANOVA

ELIGIBILITY:
Inclusion Criteria:

* • 8 to 12 years of age

  * Both male and female
  * Hemiplegic cerebral palsy according to (GMFCS) severity level I-II
  * Ability to follow instructions and participate in therapy session

Exclusion Criteria:

* • Presence of any medical conditions that would severely limit a child's participation in the study as vision or hearing loss, cardiac anomalies.

  * severe cognitive impairments that would hinder the participant's ability to actively participate in therapy sessions.
  * Complicated systemic disorders.
  * Uncontrollable seizures.
  * Usage of Botulinum toxin A injection within 3 months of prior

Ages: 8 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 32 (Actual)
Dates: Start 2023-12-01 (Actual); Primary Completion 2024-02-05 (Actual); Study Completion 2024-02-05 (Actual)

PRIMARY OUTCOMES:
Trunk Impairment Scale (TIS). | 8 weeks
  The static subscale. The dynamic subscale
  For each item, a 2-, 3- or 4-point ordinal scale is used. On the static and dynamic sitting balance and coordination subscales the maximal scores that can be attained are 7, 10 and 6 points. The total score for TIS ranges between 0 for a minimal performance to 23 for a perfect performance. In a recent version of the TIS (version 2.0) for adults, the static subscale was removed because of a ceiling effect, total score ranges between 0 and 16 points.

SECONDARY OUTCOMES:
Trunk Control Measurement Scale (TCMS). | 8 weeks
  The TCMS scale assesses seated trunk control in three dimensions. The maximum score is 58 points where 20 points correspond to static balance, 28 to selective movement control, and 10 to the ability to perform dynamic reaching TCMS sub scores appeared to be clinically relevant because children with less than around 80% of the static balance score, less than 55% of the dynamic reaching score, or less than around 35% of the selective movement control score needed support for daily life activities

CONTACTS AND LOCATIONS:
Overall Officials: Izzah Bukhtawar, MS, Principal Investigator — Riphah International University
Locations (1):
- Riphah International University, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Martins E, Cordovil R, Oliveira R, Letras S, Lourenco S, Pereira I, Ferro A, Lopes I, Silva CR, Marques M. Efficacy of suit therapy on functioning in children and adolescents with cerebral palsy: a systematic review and meta-analysis. Dev Med Child Neurol. 2016 Apr;58(4):348-60. doi: 10.1111/dmcn.12988. Epub 2015 Nov 27. PMID 26613800